CLINICAL TRIAL: NCT03753334
Title: Étude Pilote randomisée de Phase IIB, contrôlée Par placébo, évaluant l'Effet thérapeutique d'Une supplémentation en Omega-3 (Principalement EPA) Chez Des Patients en récidive Biochimique ou en Progression du Cancer de la Prostate.
Brief Title: Effects of EPA in Men With Biochemical Recurrence or Progression of Prostate Cancer.
Acronym: RCT-EPAII-BCR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-3407
Record Dates: First submitted 2018-11-14; First posted 2018-11-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Biochemical recurrence (BCR); Androgen-deprivation therapy (ADT); PSA doubling time; Quality of life; Omega-3 fatty acids; Biomarkers; Prostate cancer progression; PSA kinetics
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 1-eicosapentaenoylglycerol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAG-EPA group (Experimental): 5g/day of omega-3-rich fish oil capsules, which include 4g of purified EPA, to be taken once a day, for 12 months.
  Interventions: Combination Product: MAG-EPA
- Placebo group (Placebo Comparator): 5g/day of high-oleic sunflower oil capsules, to be taken once a day, for 12 months.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Combination Product: MAG-EPA — 5g/day of omega-3-rich fish oil including 4g of purified monoglycerides EPA, capsules, taken once daily, for 12 months
  Arms: MAG-EPA group
Dietary Supplement: Placebo group — 5g/day of placebo (high oleic sunflower oil), capsules, taken once daily, for 12 months
  Other Names: High oleic sunflower oil
  Arms: Placebo group

SUMMARY:
Prostate cancer biochemical recurrence (BCR) occurs in 20-50% of patients following radical prostatectomy or radiotherapy. Due to significant risk of side effects and uncertainty about the benefits, physicians and patients are seeking alternatives to delay androgen deprivation therapy (ADT) for non-metastatic BCR. Long-chain omega-3 fatty acids (LCn3), mainly found in seafood and fatty fish, have beneficial effects against prostate cancer in pre-clinical experimental studies and randomized clinical trials of intermediate prostate cancer outcomes. The current observational evidence also supports testing LCn3 in prostate cancer patients. LCn3 have beneficial effects on inflammation, cardiovascular, psychological, and other outcomes, contrasting sharply with ADT-associated side effects.

Investigators propose to conduct a pilot randomized placebo-controlled trial to determine the effects over one year of an innovative LCn3 supplement (5g of omega-3-rich fish oil daily, including 4g of monoglycerides eicosapentaenoic acid (MAG-EPA)) in 40 men experiencing BCR or prostate cancer progression after a curative treatment.

This project proposes a simple intervention by dietary supplementation that could eventually help to prevent or delay ADT-related side effects and thus could contribute to diminish the heavy individual and societal burden of prostate cancer. The clinical data generated by this pilot trial will serve as basis for a larger-scale phase II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed history of adenocarcinoma of the prostate.
* Patients must have a PSA failure defined as PSA of >= 0.5 ng/ml that has increased above nadir following radical prostatectomy (RP); or a PSA increase of 2.0 above post-therapy nadir after radiotherapy (RT); or a PSA increase between 0.05-0.49 ng/ml that has increased above nadir following RP. The maximal PSA value at enrolment must be <5.0 ng/mL after RP and <6 ng/mL after RT.
* PSA value must be increasing based on three consecutive measurements each separated by at least 4 weeks prior to enrolment to this study.
* Patients may have received any number of local therapies (RP, external beam RT or brachytherapy).
* Provide written informed consent.

Exclusion Criteria:

* Patients with evidence of metastatic disease.
* Patients who have received prior cytotoxic chemotherapy for recurrent disease.
* Patients currently receiving biological response modifiers, or corticosteroids.
* Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness or social situations that would limit compliance with study requirements.
* Use of omega-3 or any other dietary supplements for the previous 3 months and during study is not allowed.
* Known allergy to fish or shellfish or sunflower.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prostate-specific antigen (PSA) doubling time from baseline to 12 months. | 12 months
  Efficacy of a one-year MAG-EPA supplementation versus placebo on PSA kinetics will be evaluated based on the comparison of PSA doubling time from baseline to 12 months. The investigators will measure PSA level every three months and calculate PSA doubling time at 12 months (using a linear regression approach) after randomisation using the randomisation PSA value as the starting point. PSA slope will be defined as the linear regression line of the natural log of PSA (in ng/mL) against time (in months). PSA doubling time will be defined as the natural log of 2 divided by the PSA slope.

SECONDARY OUTCOMES:
Fatty acid profiles in red blood cells, changes relative to baseline (time 0). | 3, 6, 9,12 months
  The changes of fatty acid levels in red blood cell membranes, relative to their baseline levels, will be measured every three months. The profile of fatty acids will be quantified using gas chromatography coupled with mass spectrometry and expressed as relative percentages of total fatty acids.
Modulation of the Quality of life related to Sleep, changes relative to baseline (time 0) and between arms. | 3, 6, 9, 12 months
  The Insomnia Severity Scale (ISI, scores 0-28) and the Fatigue Symptom Inventory (FSI, scores 0-10) will be used to evaluate QoL related to sleep. For both questionnaires, higher scores mean a worse outcome.
Change in Inflammatory mediators levels | 0, 3, 12 months
  The changes in levels of systemic inflammatory mediators in both arms, relative to their baseline levels, at 3- and 12-month, will be measured. The levels of mediators will be expressed in pg/mL and quantified using validated techniques.
Modulation of the Quality of life related to Cognitive Function, changes relative to baseline (time 0) and between arms. | 3, 6, 9,12 months
  The Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) will be used to measure cognitive function. This questionnaire evaluates different subscales, i.e. Perceived Cognitive Impairments (scores 0-72), Impact of Perceived cognitive impairments (scores 0-16), Comments from Others (scores 0-16) and Perceived Cognitive Abilities (scores 0-28). For each subscale, higher scores mean a better outcome.
Modulation of the Quality of life related to Prostate Symptoms, changes relative to baseline (time 0) and between arms. | 0, 3, 6, 9, 12 months
  The International Prostate Symptom Scale (IPSS) and the Expanded Prostate Cancer Index Composite 26 (EPIC-26) will be used to measure prostate symptoms. The IPSS evaluate urinary symptoms (scores 0-35) and QoL related to these symptoms (scores 0-6). Higher scores mean a worse outcome. The EPIC-26 evaluates prostate symptoms for 5 domains (sexual, urinary incontinence, urinary irritative/obstructive, hormonal and bowel), each score ranging from 0-100. Higher scores mean a better outcome.
Modulation of the Quality of life related to Anxiety and Depression, changes relative to baseline (time 0) and between arms. | 0, 3, 6, 9, 12 months
  The Hospital Anxiety and Depression Scale (HADS) will be used to measure anxiety and depression symptoms. Both the anxiety and depression scale scores range from 0-21, where higher scores mean a worse outcome. The Patient Health Questionnaire 9 (PHQ-9, scores 0-27) will be used as well to measure depression symptoms. Higher scores mean more depressive symptoms.
Modulation of the Quality of life related to Health, changes relative to baseline (time 0) and between arms. | 0, 3, 6, 9, 12 months
  The 36-Item Short Form Health Survey (SF-36) will be used to measure health-related QoL. Scores range from 0-100 on 8 domains (physical functioning, role physical, general health, pain, social functioning, role emotional, vitality and mental health) and two component summary scales (physical and mental). Higher scores mean better health-related QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Fradet, MD, PhD, Principal Investigator — CHU de Québec-Univeristé Laval
Locations (1):
- Centre de Recherche Clinique et Évaluative en Oncologie - Hôtel-Dieu de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided